CLINICAL TRIAL: NCT03742115
Title: A Randomized Controlled Trial of Etoposide in the First-line Treatment of Adult Epstein-barr Virus Associated Hemophagocytic Lymphohistiocytosis
Brief Title: Etoposide in the First-line Treatment of Adult EBV-HLH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Dr., Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-16-adult EBV-HLH-first line
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Etoposide; Dexamethasone; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Etoposide standard group (Experimental): Etoposide 150 mg/m2 twice weekly for 2 weeks and then weekly; dexamethasone initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering
  Interventions: Drug: Etoposide; Drug: Dexamethasone
- Etoposide reduction group (Experimental): Etoposide 150 mg/m2 once a week; dexamethasone initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering
  Interventions: Drug: Dexamethasone; Drug: Etoposide
- Corticosteroid group (Active Comparator): dexamethasone initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering, with or without IvIG (0.5 g/kg IV, once every 4 weeks)
  Interventions: Drug: Dexamethasone; Drug: IVIG

INTERVENTIONS:
Drug: Etoposide — 150 mg/m2 twice weekly for 2 weeks and then weekly
  Arms: Etoposide standard group
Drug: Dexamethasone — initially 10 mg/m2 for 2 weeks followed by 5 mg/m2 for 2 weeks, 2.5 mg/m2 for 2 weeks, 1.25 mg/m2 for one week, and one week of tapering
Drug: Etoposide — 150 mg/m2 weekly
  Arms: Etoposide reduction group
Drug: IVIG — 0.5 g/kg, once every 4 weeks
  Arms: Corticosteroid group

SUMMARY:
his study aimed to investigate the efficacy of etoposide as the first line therapy for adult Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were older than 18 years of age
2. Diagnosed as EBV-Hemophagocytic Lymphohistiocytosis (HLH)
3. Patients did not receive any treatment for HLH before
4. Informed consent

Exclusion Criteria:

1. Heart function above grade II (NYHA)
2. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2
3. Pregnancy or lactating Women
4. Allergic to Pegaspargase, doxorubicin or etoposide
5. Active bleeding of the internal organs
6. uncontrollable infection
7. history of acute and chronic pancreatitis
8. Participate in other clinical research at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response(complete response+ partial response) rate of Participants | Change from before and 2,4 weeks after initiating thearpy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25(pg/ml), ferritin(μg/L), and triglyceride(mmol/L); hemoglobin(g/L); neutrophil counts(×109/L); platelet counts(×109/L); and alanine aminotransferase (ALT(U/L)).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25(pg/ml) response was>1.5-fold decreased; ferritin (μg/L)and triglyceride(mmol/L) decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT (U/L)decrease of at least 50%.

SECONDARY OUTCOMES:
Compare survival between two arms | from the time patients received therapy up to 12 months or December 2020

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 years
  Adverse events including pancreatitis, liver function damage, myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Imashuku S, Kuriyama K, Teramura T, Ishii E, Kinugawa N, Kato M, Sako M, Hibi S. Requirement for etoposide in the treatment of Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis. J Clin Oncol. 2001 May 15;19(10):2665-73. doi: 10.1200/JCO.2001.19.10.2665. PMID 11352958
- [Background] Imashuku S, Kuriyama K, Sakai R, Nakao Y, Masuda S, Yasuda N, Kawano F, Yakushijin K, Miyagawa A, Nakao T, Teramura T, Tabata Y, Morimoto A, Hibi S. Treatment of Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis (EBV-HLH) in young adults: a report from the HLH study center. Med Pediatr Oncol. 2003 Aug;41(2):103-9. doi: 10.1002/mpo.10314. PMID 12825212
- [Background] Henter JI, Samuelsson-Horne A, Arico M, Egeler RM, Elinder G, Filipovich AH, Gadner H, Imashuku S, Komp D, Ladisch S, Webb D, Janka G; Histocyte Society. Treatment of hemophagocytic lymphohistiocytosis with HLH-94 immunochemotherapy and bone marrow transplantation. Blood. 2002 Oct 1;100(7):2367-73. doi: 10.1182/blood-2002-01-0172. PMID 12239144